CLINICAL TRIAL: NCT01549730
Title: A Feasibility Study of Hypoxia Imaging in Patients With Cervix Cancer Using Positron Emission Tomography (PET) With 18F-Fluoroazomycin Arabinoside (18F-FAZA)
Brief Title: Cervix Hypoxia FAZA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UHN REB 11-0026-C
Record Dates: First submitted 2011-06-23; First posted 2012-03-09 (Estimated); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Cervix Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — fluoroazomycin arabinoside

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PET FAZA imaging (Experimental): PET FAZA imaging of tumor hypoxia in patients with cervix cancer
  Interventions: Procedure: 18F-Fluoroazomycin Arabinoside (18F-FAZA)

INTERVENTIONS:
Procedure: 18F-Fluoroazomycin Arabinoside (18F-FAZA) — A PET scan is an imaging test that uses special radioactive dyes to measure different aspects of how your cancer acts. In this study, a dye called 18F-Fluoroazomycin Arabinoside (18F-FAZA) will be used to measure hypoxia levels in tumours. Health Canada has not approved FAZA for general use, but has approved it for use in this study.

SUMMARY:
The purpose of this study is to look for low levels of oxygen (hypoxia) in your cervix cancer using a special x-ray test called a positron emission tomography (PET)scan. Hypoxia may have an effect on how cervix cancer grows and responds to treatments like radiotherapy and chemotherapy. Doctors at Princess Margaret Hospital have measured hypoxia in over 300 patients. The use of PET scans to measure hypoxia may be better and simpler than the methods used previously.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologic diagnosis of squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma of the cervix
* TNM (7th edition) cT1-4, N0-1, M0-1
* Intention to treat using radiotherapy with or without concurrent cisplatin chemotherapy according to the current treatment policies of the PMH Gynecology Group
* No cytotoxic anti-cancer therapy for cervix cancer prior to study entry
* A negative urine or serum pregnancy test within the two week interval immediately prior to PET-CT imaging, in women of child-bearing age
* Ability to provide written informed consent to participate in the study

Exclusion Criteria:

* Prior complete or partial hysterectomy
* Carcinoma of the cervical stump
* Inability to lie supine for more than 30 minutes
* Patients taking the drug disulfuram (Antabuse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of patients treated with the PET tracer FAZA to image primary tumor hypoxia in patients with cervix cancer prior to treatment with radiotherapy and concurrent cisplatin chemotherapy | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Milosevic, MD, Principal Investigator — Princess Margaret Hospital, University Health Network
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada